CLINICAL TRIAL: NCT03065517
Title: Using Mobile Technology to Enhance MST Outcomes
Brief Title: VillageWhere: Innovative Mobile Technology for Youth With Conduct Disorder and Their Parents
Acronym: VillageWhere
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evidence-Based Practice Institute, Seattle, WA (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R44MH097349 (NIH); R44MH097349 (NIH)
Record Dates: First submitted 2017-02-16; First posted 2017-02-28 (Actual); Results first posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Child Behavior Disorders
Keywords: Criminal Justice; Juvenile Delinquency
MeSH Terms: conditions — Child Behavior Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VillageWhere App (Experimental): Parent-youth dyads assigned to the VillageWhere condition will be asked to use the VillageWhere App that has been developed for this study. Parent and youth will be asked upload the app to their phone during the baseline assessment process and asked to use it as often as they would like throughout the duration of the 12 week trial. The app is designed to be used several times throughout each day.
  Interventions: Device: VillageWhere App
- Attention-Control Placebo App (Placebo Comparator): Parent-youth dyads assigned to the control condition will be asked to use a free placebo control app that is well-liked by parents and youth but void of content already part of an existing evidence-based treatment for youth with conduct problems (e.g., geolocation tracking). Parent and youth will be asked upload the app to their phone during the baseline assessment process and asked to use it as often as they would like throughout the duration of the 12 week trial.
  Interventions: Device: Attention-Control Placebo App

INTERVENTIONS:
Device: VillageWhere App — VillageWhere is a mobile phone app for use on both Android and iOS platforms by youth with conduct disorders and their parents.
  Arms: VillageWhere App
Device: Attention-Control Placebo App — Mobile phone app for use on both Android and iOS platforms.
  Arms: Attention-Control Placebo App

SUMMARY:
The goal of this Phase II Small Business Innovation Research (SBIR) is to develop, evaluate, and commercialize a linked parent-youth mobile app system, VillageWhere, to support the key treatment targets of evidence-based treatments for youth with conduct disorders: clear parental expectations, parental monitoring, discipline consistency, and parental support, while simultaneously cultivating intrinsic motivation in youth toward prosocial behaviors. When used in conjunction with an evidence-based treatment for delinquent youth, VillageWhere could help reduce treatment length and cost. When provided in non-evidence-based clinical settings, VillageWhere may increase access to state-of-the-art clinical techniques to those who might not otherwise receive them. Investigators will conduct usability and acceptability tests of new features with target-end-users (youth and their parents) and key stakeholders (i.e., probation officers, clinic administrators). Once usability and acceptability is achieved, investigators will conduct a 16-week randomized controlled trial (RCT) comparing VillageWhere to an attention-control (placebo) mobile app. We expect that across four time points, VillageWhere use will result in greater improvements in parent management practices and youth autonomy support, parent-youth communication and connectedness, youth intrinsic motivation for positive behavior, and youth conduct problems than the placebo. The RCT will occur with 100 parent-youth dyads recruited from various treatment and probation settings, and represent clinically-significant conduct-problems of various clinically-significant severity levels.

ELIGIBILITY:
Parent Inclusion Criteria:

* English speaking
* owns an Android or iPhone-based smartphone with a data plan, is the primary user of the phone, and uses it on a daily basis
* primary caregiver and has legal guardianship (custody) of a youth aged 13-18 with conduct disorder.

Parent Exclusion Criteria:

* has an open case with child protective services
* does not have legal custody of the youth
* participated in Phase I project and/or the Phase II formative evaluation

Youth Inclusion Criteria:

* English speaking
* possesses and is the primary user of an Android or iPhone-based smartphone with a data plan
* resides in the same household as the linked parent participant at least five days a week
* actively (past two weeks) engaging in clinically significant conduct-problem behaviors Note: Youth who have "stepped down" from a residential treatment or juvenile justice facility in the past month but may not have exhibited conduct problem behavior within the past 2 weeks will also be eligible, provided other criteria are met.

Youth Exclusion Criteria:

* resides with a secondary caregiver 3 or more days each week

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Dimeff, PhD, Principal Investigator — Evidence-Based Practice Institute; Cindy Schaeffer, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Evidence-Based Practice Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Requests for use of data will be considered on a case-by-case basis. Interested researchers may send data requests to research@ebpi.org.

REFERENCES:
- [Derived] Schaeffer CM, Dimeff LA, Koerner K, Chung J, Kelley-Brimer A, Kako N, Ilac M, Tuerk E, Carroll D, Beadnell B. A Smartphone App for Parental Management of Adolescent Conduct Problems: Randomized Clinical Trial of iKinnect. J Clin Child Adolesc Psychol. 2025 Jan-Feb;54(1):52-66. doi: 10.1080/15374416.2022.2070851. Epub 2022 May 31. PMID 35640058

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We received 645 dyad referrals. 40 were lost to follow-up, meaning 605 dyads completed the initial screen. 354 of those dyads were ineligible. Of the 251 dyads eligible for the study, 142 were lost to follow-up or dropped (mostly for no longer being interested) before consent. 113 dyads were consented, 110 had youth assent obtained, and 108 were randomized to a condition.
Groups:
- VillageWhere App: Parent-youth dyads assigned to the VillageWhere condition will be asked to use the VillageWhere App that has been developed for this study. Parent and youth will be asked upload the app to their phone during the baseline assessment process and asked to use it as often as they would like throughout the duration of the 16 week trial. The app is designed to be used several times throughout each day.
  VillageWhere App: VillageWhere is a mobile phone app for use on both Android and iOS platforms by youth with conduct disorders and their parents.
- Attention-Control Placebo App: Parent-youth dyads assigned to the control condition will be asked to use a free placebo control app that is well-liked by parents and youth but void of content already part of an existing evidence-based treatment for youth with conduct problems (e.g., geolocation tracking). Parent and youth will be asked upload the app to their phone during the baseline assessment process and asked to use it as often as they would like throughout the duration of the 16 week trial.
  Attention-Control Placebo App: Mobile phone app for use on both Android and iOS platforms.
Period: Overall Study
Arm/Group | VillageWhere App | Attention-Control Placebo App
Started | 110 | 106
Completed | 84 | 90
Not Completed | 26 | 16

BASELINE CHARACTERISTICS:
Population: 55 and 53 are the number of parent/youth dyads assigned to each condition.
Groups:
- Total: Total of all reporting groups
Arm/Group | VillageWhere App | Attention-Control Placebo App | Total
Number analyzed (Participants) | 55 | 53 | 108
Age, Categorical [Count of Participants; unit: Participants] — The age of the youth participating Population: Some participants have missing data (chose not to input this information).
  Participants
    number analyzed (Participants) | 50 | 51 | 101
    <=18 years | 50 | 51 | 101
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 0 | 0 | 0
Age, Categorical [Count of Participants; unit: Participants] — The age of the parents/caregivers participating
  Participants
    <=18 years | 1 | 0 | 1
    Between 18 and 65 years | 54 | 52 | 106
    >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants] — The sex of the youth participating Population: Some participants have missing data (chose not to input this information).
  Participants
    number analyzed (Participants) | 54 | 53 | 107
    Female | 25 | 23 | 48
    Male | 29 | 30 | 59
Sex: Female, Male [Count of Participants; unit: Participants] — The sex of the parents/caregivers participating
  Participants
    Female | 49 | 52 | 101
    Male | 6 | 1 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — The race/ethnicity of the parents/caregivers participating
  Participants
    Race: More than One Race or Other | 6 | 2 | 8
    Race: American Indian or Alaskan Native | 2 | 1 | 3
    Race: Asian | 1 | 1 | 2
    Race: Black | 8 | 9 | 17
    Race: White | 38 | 40 | 78
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — The race/ethnicity of the youth participating Population: Some participants have missing data (chose not to input this information).
  Participants
    Race: number analyzed (Participants) | 54 | 53 | 107
    Race: More than One Race or Other | 10 | 6 | 16
    Race: American Indian or Alaskan Native | 2 | 1 | 3
    Race: Asian | 0 | 1 | 1
    Race: Black | 10 | 10 | 20
    Race: White | 32 | 35 | 67
Region of Enrollment [Number; unit: participants] — The region of the youth participating
  participants
    United States | 55 | 53 | 108
Region of Enrollment [Number; unit: participants] — The region of the parents/caregivers participating
  participants
    United States | 55 | 53 | 108
Hispanic (Youth) [Count of Participants; unit: Participants]
  Hispanic | 15 | 5 | 20
  Not Hispanic | 40 | 48 | 88
Hispanic (Parent) [Count of Participants; unit: Participants]
  Hispanic | 46 | 3 | 49
  Not Hispanic | 9 | 50 | 59
Arrest (Youth-Only) [Count of Participants; unit: Participants] — Population: Some participants have missing data (chose not to input this information).
  Participants
    number analyzed (Participants) | 16 | 10 | 26
    Has been arrested | 7 | 5 | 12
    Has not been arrested | 9 | 5 | 14
Education (Youth) [Count of Participants; unit: Participants] — Population: Some participants have missing data (chose not to input this information).
  Participants
    number analyzed (Participants) | 54 | 53 | 107
    Completed 6th grade | 7 | 3 | 10
    Completed 7th grade | 9 | 11 | 20
    Completed 8th grade | 13 | 9 | 22
    Completed 9th grade | 14 | 14 | 28
    Completed 10th grade | 5 | 11 | 16
    Completed 11th grade | 5 | 2 | 7
    High school graduate | 1 | 1 | 2
    Completed 5th grade | 0 | 2 | 2
Education (Parent) [Count of Participants; unit: Participants]
  Other | 7 | 1 | 8
  Completed 9th grade | 0 | 2 | 2
  Completed 10th grade | 2 | 1 | 3
  High school graduate | 18 | 25 | 43
  2-year college degree | 10 | 9 | 19
  4-year college degree | 15 | 9 | 24
  4-year degree + Masters | 2 | 5 | 7
  PhD, MD, or other doctoral degree | 1 | 1 | 2
Relationship Status (Parent-only) [Count of Participants; unit: Participants]
  Other | 3 | 3 | 6
  Single | 12 | 14 | 26
  Single and living with my partner | 5 | 9 | 14
  Married and living with teens parent | 18 | 15 | 33
  Married and living with someone other than teens parent | 5 | 10 | 15
  Separated or divorced/divorcing from the teens parent | 10 | 0 | 10
  Separated or divorced/divorcing from someone other than the teens parent | 2 | 2 | 4
Relationship to Teen (Parent-only) [Count of Participants; unit: Participants]
  Biological Parent | 49 | 46 | 95
  Adoptive Parent | 4 | 3 | 7
  Stepparent | 1 | 1 | 2
  Grandparent | 1 | 1 | 2
  Family Member Other Than Parent | 0 | 1 | 1
  Other | 0 | 1 | 1
Employment (Parent-only) [Count of Participants; unit: Participants] — Population: Some participants have missing data (chose not to input this information).
  Participants
    number analyzed (Participants) | 55 | 52 | 107
    Employed | 31 | 38 | 69
    Unemployed | 24 | 14 | 38
Income (Parent-only) [Count of Participants; unit: Participants]
  Less than $10,000 | 7 | 6 | 13
  $10,001 to $20,000 | 8 | 6 | 14
  $20,001 to $30,000 | 6 | 13 | 19
  $30,001 to $40,000 | 6 | 4 | 10
  $40,001 to $50,000 | 4 | 5 | 9
  $50,001 to $60,000 | 7 | 7 | 14
  $60,000 and above | 17 | 12 | 29

OUTCOME MEASURES:

1. Primary Outcome: Child Behavior Checklist (CBCL)
Description: Assesses parent report of youth rule-breaking, aggressive, anxious/depressed, and drug/alcohol use behaviors. Contains two subscales: rule-breaking (minimum of 0, maximum of 36) and aggressive behavior (minimum of 0, maximum of 34). Higher scores are a worse outcome.
Time Frame: Baseline (time 1), 4-week follow-up (time 2), 8-week follow-up (time 3), and 12-week follow-up (time 4).
Population: The number analyzed differs between rows because of attrition over different timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VillageWhere App | Attention-Control Placebo App
Number analyzed (Participants) | 55 | 53
score on a scale
  Rule-Breaking Time 1 | 10.73 (5.86) | 11.45 (5.51)
  Rule-Breaking Time 2: number analyzed (Participants) | 42 | 45
  Rule-Breaking Time 2 | 7.88 (5.50) | 7.49 (5.19)
  Rule-Breaking Time 3: number analyzed (Participants) | 42 | 45
  Rule-Breaking Time 3 | 6.98 (5.43) | 7.31 (5.90)
  Rule-Breaking Time 4: number analyzed (Participants) | 41 | 44
  Rule-Breaking Time 4 | 7.12 (5.95) | 6.69 (6.29)
  Aggressive Behavior Time 1 | 19.31 (8.22) | 20.53 (7.80)
  Aggressive Behavior Time 2: number analyzed (Participants) | 42 | 45
  Aggressive Behavior Time 2 | 14.14 (6.43) | 13.53 (7.84)
  Aggressive Behavior Time 3: number analyzed (Participants) | 42 | 45
  Aggressive Behavior Time 3 | 11.93 (7.40) | 12.89 (7.50)
  Aggressive Behavior Time 4: number analyzed (Participants) | 41 | 44
  Aggressive Behavior Time 4 | 10.93 (8.23) | 12.70 (8.48)

2. Primary Outcome: Youth Self-Report (YSR)
Description: Assesses youth self-report of rule-breaking, aggressive, anxious/depressed, and drug/alcohol use behaviors. Contains two subscales: rule-breaking (minimum of 0, maximum of 34) and aggressive behavior (minimum of 0, maximum of 36). Higher scores indicate worse outcomes.
Time Frame: Baseline (time 1), 4-week follow-up (time 2), 8-week follow-up (time 3), and 12-week follow-up (time 4).
Population: The number analyzed differs between rows because of attrition over timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VillageWhere App | Attention-Control Placebo App
Number analyzed (Participants) | 55 | 52
score on a scale
  Rule-Breaking Time 1 | 11.07 (5.66) | 10.33 (4.87)
  Rule-Breaking Time 2: number analyzed (Participants) | 41 | 45
  Rule-Breaking Time 2 | 9.41 (4.38) | 8.40 (4.34)
  Rule-Breaking Time 3: number analyzed (Participants) | 40 | 43
  Rule-Breaking Time 3 | 9.50 (5.41) | 7.02 (3.38)
  Rule-Breaking Time 4: number analyzed (Participants) | 40 | 41
  Rule-Breaking Time 4 | 9.70 (5.38) | 7.07 (4.71)
  Aggressive Behavior Time 1 | 16.22 (7.50) | 15.25 (7.05)
  Aggressive Behavior Time 2: number analyzed (Participants) | 41 | 45
  Aggressive Behavior Time 2 | 13.88 (6.54) | 11.86 (5.79)
  Aggressive Behavior Time 3: number analyzed (Participants) | 40 | 43
  Aggressive Behavior Time 3 | 12.08 (6.60) | 9.67 (5.29)
  Aggressive Behavior Time 4: number analyzed (Participants) | 40 | 41
  Aggressive Behavior Time 4 | 11.93 (8.40) | 10.51 (5.86)

3. Primary Outcome: Self-Report of Delinquent Behavior Scale
Description: Assesses youth delinquent behaviors. Contains one main scale: the general delinquency scale. There are also several subscales: the status offenses (e.g., ran away from home, purchased alcohol, truant) subscale, the school delinquency subscale (e.g., cheated on tests, damaged school property, got suspended), the minor theft subscale, and the robbery subscale. For all scales, participants reported the number of times in the past two weeks they did a variety of actions; scales were then calculated as the sum of the occurrences. The minimum of each scale was 0 and there was no maximum, since there is no maximum amount participants could have done the actions listed.
Time Frame: Baseline (time 1), 4-week follow-up (time 2), 8-week follow-up (time 3), and 12-week follow-up (time 4).
Population: Number analyzed differs between rows because of attrition over timepoints.
Measure: Mean (Standard Deviation); unit: Occurrences
Arm/Group | VillageWhere App | Attention-Control Placebo App
Number analyzed (Participants) | 55 | 51
Occurrences
  General Delinquency Time 1 | 16.91 (64.41) | 7.96 (14.0)
  General Delinquency Time 2: number analyzed (Participants) | 40 | 45
  General Delinquency Time 2 | 9.03 (15.80) | 4.29 (10.14)
  General Delinquency Time 3: number analyzed (Participants) | 39 | 43
  General Delinquency Time 3 | 3.74 (5.87) | 3.98 (10.12)
  General Delinquency Time 4: number analyzed (Participants) | 37 | 41
  General Delinquency Time 4 | 2.97 (4.73) | 3.32 (5.52)
  Status Offenses Time 1: number analyzed (Participants) | 53 | 51
  Status Offenses Time 1 | 3.04 (11.13) | 2.24 (3.97)
  Status Offenses Time 2: number analyzed (Participants) | 40 | 45
  Status Offenses Time 2 | .9 (1.66) | .67 (1.28)
  Status Offenses Time 3: number analyzed (Participants) | 39 | 42
  Status Offenses Time 3 | 0.74 (1.74) | 1.04 (2.25)
  Status Offenses Time 4: number analyzed (Participants) | 37 | 41
  Status Offenses Time 4 | .73 (1.91) | 1.15 (2.74)
  School Delinquency Time 1: number analyzed (Participants) | 54 | 51
  School Delinquency Time 1 | 6.24 (21.56) | 3.41 (5.71)
  School Delinquency Time 2: number analyzed (Participants) | 40 | 45
  School Delinquency Time 2 | 5.18 (10.83) | 1.8 (4.72)
  School Delinquency Time 3: number analyzed (Participants) | 39 | 43
  School Delinquency Time 3 | 1.72 (3.62) | 1.64 (3.61)
  School Delinquency Time 4: number analyzed (Participants) | 37 | 41
  School Delinquency Time 4 | 1.41 (2.80) | 1.39 (2.87)
  Minor Theft Time 1 | 0 (0) | 0 (0)
  Minor Theft Time 2: number analyzed (Participants) | 40 | 45
  Minor Theft Time 2 | 0 (0) | 0 (0)
  Minor Theft Time 3: number analyzed (Participants) | 39 | 43
  Minor Theft Time 3 | 0 (0) | 0 (0)
  Minor Theft Time 4: number analyzed (Participants) | 37 | 41
  Minor Theft Time 4 | 0 (0) | 0 (0)
  Robbery Time 1 | 0 (0) | 0 (0)
  Robbery Time 2: number analyzed (Participants) | 40 | 45
  Robbery Time 2 | 0 (0) | 0 (0)
  Robbery Time 3: number analyzed (Participants) | 39 | 43
  Robbery Time 3 | 0 (0) | 0 (0)
  Robbery Time 4: number analyzed (Participants) | 37 | 41
  Robbery Time 4 | 0 (0) | 0 (0)

4. Primary Outcome: GAIN Substance Frequency Scale
Description: The Global Appraisal of Individual Needs (GAIN) substance frequency scale assesses youth alcohol and substance use in the last two weeks. Alcohol days are number of days in the past two weeks that youth consumed alcohol. Drunk days are the number of days in the past two weeks that youth were drunk. Marijuana days are number of days in the past two weeks that youth used marijuana. As such, the minimum and maximum values are 0 and 14, respectively, and higher scores mean a worse outcome.
Time Frame: Baseline (time 1), 4-week follow-up (time 2), 8-week follow-up (time 3), and 12-week follow-up (time 4).
Population: Number analyzed differs between rows because of attrition over timepoints.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | VillageWhere App | Attention-Control Placebo App
Number analyzed (Participants) | 55 | 52
Days
  Alcohol Days Time 1 | .76 (2.227) | .48 (1.488)
  Alcohol Days Time 2: number analyzed (Participants) | 41 | 45
  Alcohol Days Time 2 | .15 (.573) | .00 (.00)
  Alcohol Days Time 3: number analyzed (Participants) | 40 | 43
  Alcohol Days Time 3 | .30 (.791) | .23 (.782)
  Alcohol Days Time 4: number analyzed (Participants) | 40 | 41
  Alcohol Days Time 4 | .25 (.776) | .12 (.640)
  Drunk Days Time 1 | .51 (1.999) | .17 (.734)
  Drunk Days Time 2: number analyzed (Participants) | 41 | 45
  Drunk Days Time 2 | .00 (.00) | .00 (.00)
  Drunk Days Time 3: number analyzed (Participants) | 40 | 43
  Drunk Days Time 3 | .18 (.594) | .16 (.531)
  Drunk Days Time 4: number analyzed (Participants) | 40 | 41
  Drunk Days Time 4 | .05 (.316) | .34 (1.353)
  Marijuana Days Time 1: number analyzed (Participants) | 54 | 52
  Marijuana Days Time 1 | 1.63 (3.808) | 1.50 (4.152)
  Marijuana Days Time 2: number analyzed (Participants) | 41 | 45
  Marijuana Days Time 2 | .54 (1.951) | 1.13 (3.307)
  Marijuana Days Time 3: number analyzed (Participants) | 40 | 43
  Marijuana Days Time 3 | 1.25 (2.976) | 1.47 (3.832)
  Marijuana Days Time 4: number analyzed (Participants) | 40 | 41
  Marijuana Days Time 4 | .80 (2.544) | 1.12 (3.716)

5. Primary Outcome: Intrinsic Motivation Inventory (IMI) Perceived Competence Scale (PCS)
Description: Assesses youth intrinsic motivation for prosocial behaviors. Contains four subscales: interest/enjoyment (minimum of 7, maximum of 49), perceived competence (minimum of 6, maximum of 42), value/usefulness (minimum of 7, maximum of 49), and effort/importance (minimum of 5, maximum of 35).
Time Frame: Baseline (time 1), 4-week follow-up (time 2), 8-week follow-up (time 3), and 12-week follow-up (time 4).
Population: Number analyzed differs between rows because of attrition over timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VillageWhere App | Attention-Control Placebo App
Number analyzed (Participants) | 55 | 52
score on a scale
  Interest/Enjoyment Time 1 | 18.54 (7.71) | 22.27 (9.18)
  Interest/Enjoyment Time 2: number analyzed (Participants) | 41 | 45
  Interest/Enjoyment Time 2 | 20.68 (7.00) | 24.00 (6.80)
  Interest/Enjoyment Time 3: number analyzed (Participants) | 40 | 43
  Interest/Enjoyment Time 3 | 21.60 (8.96) | 24.21 (10.62)
  Interest/Enjoyment Time 4: number analyzed (Participants) | 38 | 41
  Interest/Enjoyment Time 4 | 22.74 (6.20) | 23.71 (8.31)
  Perceived Competence Time 1 | 24.20 (9.64) | 23.90 (8.78)
  Perceived Competence Time 2: number analyzed (Participants) | 41 | 45
  Perceived Competence Time 2 | 25.32 (6.20) | 25.69 (7.43)
  Perceived Competence Time 3: number analyzed (Participants) | 40 | 42
  Perceived Competence Time 3 | 23.88 (7.21) | 27.38 (8.66)
  Perceived Competence Time 4: number analyzed (Participants) | 38 | 41
  Perceived Competence Time 4 | 27.66 (6.95) | 26.76 (8.71)
  Value/Usefulness Time 1 | 27.91 (12.06) | 32.40 (11.92)
  Value/Usefulness Time 2: number analyzed (Participants) | 41 | 45
  Value/Usefulness Time 2 | 28.80 (8.74) | 31.96 (9.90)
  Value/Usefulness Time 3: number analyzed (Participants) | 40 | 43
  Value/Usefulness Time 3 | 27.23 (10.30) | 31.88 (11.27)
  Value/Usefulness Time 4: number analyzed (Participants) | 38 | 41
  Value/Usefulness Time 4 | 30.05 (9.55) | 31.95 (10.05)
  Effort/Importance Time 1 | 19.15 (4.93) | 20.19 (4.91)
  Effort/Importance Time 2: number analyzed (Participants) | 41 | 45
  Effort/Importance Time 2 | 18.95 (3.71) | 21.56 (5.01)
  Effort/Importance Time 3: number analyzed (Participants) | 40 | 43
  Effort/Importance Time 3 | 19.48 (4.60) | 21.81 (4.61)
  Effort/Importance Time 4: number analyzed (Participants) | 38 | 41
  Effort/Importance Time 4 | 19.68 (3.76) | 20.39 (3.91)

6. Primary Outcome: Perceived Autonomy Support (PAS)
Description: Assesses youth perceived autonomy-supportive and controlling parent behaviors. Contains four subscales: autonomy support, chaos, coercion, and structure. Each subscale has a youth version (minimum 4, maximum 16) and a parent version (minimum 5, maximum 20). Higher scores indicate better outcomes on the autonomy and structure scales and worse outcomes on the chaos and coercion scales.
Time Frame: Baseline (time 1), 4-week follow-up (time 2), 8-week follow-up (time 3), and 12-week follow-up (time 4).
Population: Number analyzed in rows differs from overall number analyzed because of separation of youth and parent subscales and attrition over timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VillageWhere App | Attention-Control Placebo App
Number analyzed (Participants) | 108 | 105
score on a scale
  Parent Autonomy Time 1: number analyzed (Participants) | 54 | 53
  Parent Autonomy Time 1 | 15.20 (3.07) | 15.23 (3.17)
  Parent Autonomy Time 2: number analyzed (Participants) | 42 | 45
  Parent Autonomy Time 2 | 15.33 (2.67) | 15.71 (2.87)
  Parent Autonomy Time 3: number analyzed (Participants) | 41 | 45
  Parent Autonomy Time 3 | 15.46 (2.99) | 15.98 (2.90)
  Parent Autonomy Time 4: number analyzed (Participants) | 41 | 44
  Parent Autonomy Time 4 | 16.20 (2.84) | 15.98 (3.30)
  Parent Chaos Time 1: number analyzed (Participants) | 54 | 53
  Parent Chaos Time 1 | 8.20 (2.59) | 7.91 (2.43)
  Parent Chaos Time 2: number analyzed (Participants) | 42 | 45
  Parent Chaos Time 2 | 7.83 (2.61) | 8.24 (3.61)
  Parent Chaos Time 3: number analyzed (Participants) | 41 | 45
  Parent Chaos Time 3 | 8.10 (2.54) | 7.76 (3.08)
  Parent Chaos Time 4: number analyzed (Participants) | 41 | 44
  Parent Chaos Time 4 | 7.22 (2.04) | 7.91 (3.83)
  Parent Coercion Time 1: number analyzed (Participants) | 54 | 53
  Parent Coercion Time 1 | 13.22 (3.63) | 12.81 (3.83)
  Parent Coercion Time 2: number analyzed (Participants) | 42 | 45
  Parent Coercion Time 2 | 12.00 (3.38) | 11.78 (3.62)
  Parent Coercion Time 3: number analyzed (Participants) | 41 | 45
  Parent Coercion Time 3 | 12.00 (3.22) | 11.62 (3.77)
  Parent Coercion Time 4: number analyzed (Participants) | 41 | 44
  Parent Coercion Time 4 | 11.46 (3.44) | 10.89 (3.94)
  Parent Structure Time 1: number analyzed (Participants) | 54 | 53
  Parent Structure Time 1 | 16.35 (2.70) | 16.17 (3.37)
  Parent Structure Time 2: number analyzed (Participants) | 42 | 45
  Parent Structure Time 2 | 16.17 (2.68) | 16.24 (2.91)
  Parent Structure Time 3: number analyzed (Participants) | 41 | 45
  Parent Structure Time 3 | 16.85 (2.47) | 17.11 (2.96)
  Parent Structure Time 4: number analyzed (Participants) | 41 | 44
  Parent Structure Time 4 | 17.46 (2.65) | 16.80 (3.40)
  Youth Autonomy Time 1: number analyzed (Participants) | 54 | 52
  Youth Autonomy Time 1 | 9.48 (3.25) | 10.48 (3.37)
  Youth Autonomy Time 2: number analyzed (Participants) | 41 | 45
  Youth Autonomy Time 2 | 9.46 (2.65) | 9.98 (3.49)
  Youth Autonomy Time 3: number analyzed (Participants) | 40 | 43
  Youth Autonomy Time 3 | 9.60 (3.12) | 10.47 (2.82)
  Youth Autonomy Time 4: number analyzed (Participants) | 39 | 41
  Youth Autonomy Time 4 | 9.69 (3.05) | 10.78 (3.31)
  Youth Chaos Time 1: number analyzed (Participants) | 54 | 52
  Youth Chaos Time 1 | 8.11 (3.15) | 8.52 (2.94)
  Youth Chaos Time 2: number analyzed (Participants) | 41 | 45
  Youth Chaos Time 2 | 8.10 (2.96) | 8.42 (2.84)
  Youth Chaos Time 3: number analyzed (Participants) | 40 | 43
  Youth Chaos Time 3 | 8.23 (3.03) | 7.67 (2.96)
  Youth Chaos Time 4: number analyzed (Participants) | 39 | 41
  Youth Chaos Time 4 | 8.30 (3.20) | 8.24 (3.35)
  Youth Coercion Time 1: number analyzed (Participants) | 54 | 52
  Youth Coercion Time 1 | 9.93 (2.52) | 10.10 (2.54)
  Youth Coercion Time 2: number analyzed (Participants) | 41 | 45
  Youth Coercion Time 2 | 9.56 (2.61) | 9.58 (2.48)
  Youth Coercion Time 3: number analyzed (Participants) | 40 | 43
  Youth Coercion Time 3 | 9.65 (2.32) | 9.30 (2.44)
  Youth Coercion Time 4: number analyzed (Participants) | 39 | 41
  Youth Coercion Time 4 | 9.46 (2.76) | 9.39 (2.65)
  Youth Structure Time 1: number analyzed (Participants) | 54 | 52
  Youth Structure Time 1 | 10.46 (3.33) | 11.35 (3.17)
  Youth Structure Time 2: number analyzed (Participants) | 41 | 45
  Youth Structure Time 2 | 10.02 (3.08) | 10.44 (3.33)
  Youth Structure Time 3: number analyzed (Participants) | 40 | 43
  Youth Structure Time 3 | 10.05 (3.10) | 10.67 (3.15)
  Youth Structure Time 4: number analyzed (Participants) | 39 | 41
  Youth Structure Time 4 | 9.83 (3.20) | 10.37 (3.37)

7. Primary Outcome: Perceived Stress Scale (PSS)
Description: Assesses parent perception of life stress. Minimum value is 0, maximum value is 40. Higher scores mean a worse outcome.
Time Frame: Baseline (time 1), 4-week follow-up (time 2), 8-week follow-up (time 3), and 12-week follow-up (time 4).
Population: The number analyzed differs in the rows because of attrition over time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VillageWhere App | Attention-Control Placebo App
Number analyzed (Participants) | 54 | 53
score on a scale
  Time 1 | 22.06 (7.29) | 20.74 (5.34)
  Time 2: number analyzed (Participants) | 42 | 45
  Time 2 | 18.83 (5.56) | 19.62 (5.99)
  Time 3: number analyzed (Participants) | 41 | 45
  Time 3 | 18.61 (7.70) | 18.56 (6.51)
  Time 4: number analyzed (Participants) | 41 | 44
  Time 4 | 16.68 (8.06) | 17.45 (5.70)

8. Primary Outcome: Parent Locus of Control Scale
Description: Assesses parent sense of control/efficacy and supervision of youth. One sub-scale for helplessness and one sub-scale for feeling out of control. Both subscales have a minimum of 10 and maximum of 50. Higher scores are a worse outcome.
Time Frame: Baseline (time 1), 4-week follow-up (time 2), 8-week follow-up (time 3), and 12-week follow-up (time 4).
Population: Number analyzed in certain rows differs from overall number analyzed because of attrition over timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VillageWhere App | Attention-Control Placebo App
Number analyzed (Participants) | 55 | 53
score on a scale
  Helpless Time 1 | 24.80 (5.40) | 24.77 (5.37)
  Helpless Time 2: number analyzed (Participants) | 42 | 45
  Helpless Time 2 | 22.67 (4.30) | 22.71 (4.98)
  Helpless Time 3: number analyzed (Participants) | 41 | 45
  Helpless Time 3 | 22.73 (4.31) | 22.40 (6.15)
  Helpless Time 4: number analyzed (Participants) | 41 | 44
  Helpless Time 4 | 21.29 (5.22) | 21.14 (5.33)
  Out of Control Time 1 | 32.84 (7.85) | 34.23 (7.13)
  Out of Control Time 2: number analyzed (Participants) | 42 | 45
  Out of Control Time 2 | 31.31 (6.56) | 30.53 (7.95)
  Out of Control Time 3: number analyzed (Participants) | 41 | 45
  Out of Control Time 3 | 29.78 (6.60) | 29.33 (9.26)
  Out of Control Time 4: number analyzed (Participants) | 41 | 44
  Out of Control Time 4 | 27.49 (8.00) | 27.93 (8.97)

9. Primary Outcome: Loeber Parenting Scale
Description: Assesses parent and youth clarity of expectations, discipline consistency/effectiveness, and use of rewards. Subscales are Supervision (minimum of 10 and a maximum of 28 for both the parent and youth scales), Inconsistent Discipline (minimum of 9 and a maximum of 27 for the youth scale, minimum of 5 and maximum of 15 for the parent scales), Reward Use (minimum of 9 and maximum of 27 for both parent and youth scales), and Discipline Effectiveness (minimum of 3 and a maximum of 10 on the parents scale, no youth scale); higher scores mean higher prevalence, lower scores mean infrequency.
Time Frame: Baseline (time 1), 4-week follow-up (time 2), 8-week follow-up (time 3), and 12-week follow-up (time 4).
Population: The number analyzed differs between rows because of attrition over timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | VillageWhere App | Attention-Control Placebo App
Number analyzed (Participants) | 54 | 53
score on a scale
  Supervision Time 1 | 26.33 (3.08) | 25.53 (3.69)
  Supervision Time 2: number analyzed (Participants) | 42 | 45
  Supervision Time 2 | 21.98 (1.70) | 22.04 (2.14)
  Supervision Time 3: number analyzed (Participants) | 41 | 45
  Supervision Time 3 | 22.00 (1.91) | 22.53 (2.14)
  Supervision Time 4: number analyzed (Participants) | 41 | 44
  Supervision Time 4 | 22.44 (1.87) | 22.23 (2.26)
  Inconsistent Discipline Time 1 | 8.40 (2.02) | 8.43 (2.27)
  Inconsistent Discipline Time 2: number analyzed (Participants) | 42 | 45
  Inconsistent Discipline Time 2 | 7.50 (1.85) | 7.80 (2.16)
  Inconsistent Discipline Time 3: number analyzed (Participants) | 41 | 45
  Inconsistent Discipline Time 3 | 7.71 (2.00) | 7.98 (2.37)
  Inconsistent Discipline Time 4: number analyzed (Participants) | 41 | 44
  Inconsistent Discipline Time 4 | 7.02 (1.80) | 7.82 (2.34)
  Reward Use Time 1 | 21.09 (2.47) | 21.19 (3.43)
  Reward Use Time 2: number analyzed (Participants) | 42 | 45
  Reward Use Time 2 | 21.50 (2.81) | 21.87 (3.00)
  Reward Use Time 3: number analyzed (Participants) | 41 | 44
  Reward Use Time 3 | 21.90 (2.53) | 21.87 (3.14)
  Reward Use Time 4: number analyzed (Participants) | 41 | 44
  Reward Use Time 4 | 22.22 (2.58) | 21.68 (2.77)
  Discipline Effectiveness Time 1 | 5.94 (1.86) | 5.77 (1.90)
  Discipline Effectiveness Time 2: number analyzed (Participants) | 42 | 45
  Discipline Effectiveness Time 2 | 6.60 (1.71) | 6.69 (2.16)
  Discipline Effectiveness Time 3: number analyzed (Participants) | 41 | 45
  Discipline Effectiveness Time 3 | 6.73 (1.63) | 6.93 (2.19)
  Discipline Effectiveness Time 4: number analyzed (Participants) | 41 | 44
  Discipline Effectiveness Time 4 | 7.22 (1.84) | 7.23 (2.21)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Participants were asked to report potential and actual adverse events, whether or not the individual considered the event resulting from the research, via online survey, to IRB, or study PI.
Arm/Group | VillageWhere App | Attention-Control Placebo App
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/106
Serious Adverse Events (participants affected / at risk) | 0/110 | 0/106
Other Adverse Events (participants affected / at risk) | 0/110 | 0/106

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT03065517/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-29): https://cdn.clinicaltrials.gov/large-docs/17/NCT03065517/ICF_001.pdf